CLINICAL TRIAL: NCT00732108
Title: Efficacy of Topiramate in Patients Wih Migraine-Associated Dizziness
Brief Title: Is Topiramate Effective in Treating Dizziness in Patient's With Migraine-Associated Dizziness
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects enrolled
Sponsor: University of California, San Francisco (Other)
Collaborators: American Academy of Otolaryngology-Head and Neck Surgery Foundation (Other)
Responsible Party: Lawrence R. Lustig, M.D., University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H48626-32352-01
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Migraine; Headache; Dizziness
Keywords: migraine; headache; dizziness; vertigo; topiramate; Topamax
MeSH Terms: conditions — Migraine Disorders; Headache; Dizziness; Vertigo | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- topiramate (Experimental): topiramate 50mg orally for 2 weeks, then 100mg orally for 6 weeks
  Interventions: Drug: topiramate
- 2 (Placebo Comparator): 1 placebo pill orally for 2 weeks, then 2 placebo pills orally for 6 weeks
  Interventions: Drug: lactulose placebo pill

INTERVENTIONS:
Drug: topiramate — 50mg orally for 2 weeks, then 100mg orally for 6 weeks
  Other Names: Topamax
  Arms: topiramate
Drug: lactulose placebo pill — 1 placebo pill orally for 2 weeks, then 2 placebo pills orally for 6 weeks
  Other Names: placebo pill
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether topiramate effective in treating dizziness symptoms that are associated with migraine headaches.

DETAILED DESCRIPTION:
Migraine is a common disorder, often associated with dizziness symptoms. In many cases, dizziness is one of the only manifestations of migraine headaches. Various classes of drugs have been advocated as treatment for migraine-associated dizziness, though none has been shown to be superior over the others.

Topiramate is a drug approved for migraine prophylaxis. This study is designed to assess if there are significant changes in dizziness frequency and severity in patients diagnosed with migraine-associated dizziness treated with topiramate. Demonstrating benefit of topiramate with a placebo-controlled study to alleviate symptoms of dizziness would serve to clarify effective treatment options for patients with migraine-associated dizziness.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of migraine-associated dizziness.

Exclusion Criteria:

* Previous or current use of topiramate prior to study enrollment.
* Need for continued use of the following medications for any medical reason during the study: ergots, anti-epileptics, beta-blockers, calcium channel blockers, monoamine oxidase inhibitors, high-dose magnesium, high-dose riboflavin, corticosteroids, local anesthetics, botulinum toxin, or herbal preparations.
* History of nephrolithiasis.
* Women whom are pregnant or breastfeeding.
* Patients with known sensitivity to topiramate.
* Patients with a history of glaucoma.
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Change in mean 28-day monthly vertigo frequency from baseline. | 4 weeks, 8 weeks
Change in Dizziness Handicap Inventory scores from baseline. | 4 weeks, 8 weeks

SECONDARY OUTCOMES:
Change in an individual's perception of vertigo symptoms based on a 1 to 10 scale. | 4 weeks, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence R Lustig, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States